CLINICAL TRIAL: NCT02889289
Title: Balance and Endurance Outcomes for Chronic TBI Using the Xbox Kinect
Brief Title: Using the Xbox Kinect for Chronic TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01729
Record Dates: First submitted 2016-06-28; First posted 2016-09-05 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2016-10

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; virtual reality; Xbox kinect; balance
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Xbox One Kinect Gaming (Experimental): 15 sessions of supervised physical therapy using 2 commercially available Xbox One Kinect game.
  Interventions: Other: Xbox One Kinect Gaming

INTERVENTIONS:
Other: Xbox One Kinect Gaming — The Veteran completed 15 sessions of supervised VR training. Each session lasted between 50 and 60 minutes in total. The intervention utilized 2 commercially available Xbox One Kinect games called "Shape Up" and "Kinect Sports: Rivals" to challenge both cardiovascular and balance systems. Each game is composed of mini-games (MG). Each MG lasted between 1:30 minutes to 4:00 minutes. Both games were played for approximately 25 minutes during each session. Rest breaks were allowed as the participant required them. Guarding by a therapist was provided dependent on the challenge of the game and the participant's abilities.

SUMMARY:
This study will evaluate the potential for improving balance for a single individual with a history of traumatic brain injury (TBI). The participant will engage in supervised therapy using commercial games on the Xbox Kinect. This study will also evaluate the viability of improving cardiovascular fitness using this intervention as well. The investigators hypothesize that balance improvements will occur and that using the Xbox Kinect is a viable way of improving cardiovascular fitness.

DETAILED DESCRIPTION:
Various forms of virtual reality (VR) training have been recently used for rehabilitation of neurological impairments including postural stability and coordination. Virtual reality training has also been shown to increase motivation and attention through its use of novel goal-directed challenges. The Xbox Kinect gaming system allows the Veteran to perform challenging full-body and goal-oriented activities. Balance improvements using laboratory developed games have been demonstrated in those with a history of TBI. However, the investigators are specifically interested if improvements can be made using commercial games which can be utilized in physical therapy clinics more readily. Exercise gaming has been shown to provide adequate intensity exercise to improve heart health in the healthy population. However, such benefits have not yet been investigated using the Xbox Kinect for individuals with a history of TBI.

ELIGIBILITY:
Inclusion Criteria:

* A male or female Veteran participant must have sustained traumatic brain injury greater than 1 year prior to baseline assessments
* Veteran will be between the ages of 18 and 65 years old

Exclusion Criteria:

* Veterans with any cardiac condition that may cause sudden decompensation during cardiovascular testing and training (e.g., severe congestive heart failure and uncontrolled hypertension)
* If Veteran has a significant cardiac history (as defined by American College of Sports Medicine), physician approval will be acquired prior to cardiac stress tests
* Veterans with a previous history of behavioral impairments (e.g., aggression or inappropriate actions) that would preclude participation in standard physical therapy
* Veterans with lower extremity amputation
* Veterans that exhibit greater than mild cognitive impairments as shown by a score 17/30 or less on the Montreal Cognitive Assessment (MoCA).
* Veterans that are unable to stand unsupported for at least 2 minutes
* Veterans that are unable to ambulate on treadmill with bilateral hand support

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chanpimol S, Seamon B, Hernandez H, Harris-Love M, Blackman MR. Using Xbox kinect motion capture technology to improve clinical rehabilitation outcomes for balance and cardiovascular health in an individual with chronic TBI. Arch Physiother. 2017;7:6. doi: 10.1186/s40945-017-0033-9. Epub 2017 May 31. PMID 28824816

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One Veteran recruited from Polytrauma department of Washington DC VA Medical Center during April 2015.
Period: Overall Study
Arm/Group | Xbox One Kinect Gaming
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Dynamic Gait Index (DGI)
Description: The DGI is a common clinical measure used to evaluate dynamic balance and coordination during a person's daily activities. This test was developed by Shumway-Cook and features 8-items which assess a person's ability to walk while turning their head, changing speed, and navigating obstacles. The DGI is scored from 0 to 24 where higher scores indicate higher dynamic balance function.
Time Frame: Changes from (Baseline) Weeks 1,2,3,4,6,13,14 to (Intervention) Weeks 1, 3, 4, 6, 8 and to (Retention) Weeks 1, 2, 3, 4, 5
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
units on a scale
  Baseline | 12 (0.38)
  Intervention | 17 (2.28)
  Retention | 19 (0)

2. Secondary Outcome: Limits of Stability (LOS) - Directional Control
Description: The LOS is performed on the NeuroCom Balance Manager. The LOS test is a goal-directed weight shifting task. The LOS-directional control measures the accuracy of an individual's movement of center of gravity during the task compared to a straight line. This is reported as a percentage without units.
Time Frame: (Baseline) Weeks 1,2,3,4,6,13,14; (Intervention) Weeks 1, 3, 4, 6, 8; (Retention) Weeks 1, 2, 3, 4, 5
Measure: Median (Standard Deviation); unit: percentage of accuracy
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
percentage of accuracy
  Baseline | 65 (4.64)
  Intervention | 68 (3.77)
  Retention | 67 (2.19)

3. Secondary Outcome: Heart Rate at End of Mini-game
Description: Heart rated recorded using heart monitor and chest strap at the end of each mini-game.
Time Frame: (Intervention) 2 times per week for 8 weeks
Measure: Mean (Standard Deviation); unit: Heart beats per minute
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
Heart beats per minute
  1st 5 Interventions | 109.13 (12.65)
  2nd 5 interventions | 102.09 (5.78)
  3rd 5 interventions | 92.87 (3.07)

4. Secondary Outcome: Heart Rate at Beginning of Mini-game
Description: Heart rated recorded using heart monitor and chest strap at the beginning of each mini-game.
Time Frame: (Intervention) 2 times per week for 8 weeks
Measure: Mean (Standard Deviation); unit: Heart beats per minute
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
Heart beats per minute
  1st 5 Interventions | 90.71 (13.41)
  2nd 5 interventions | 87.79 (6.80)
  3rd 5 interventions | 77.95 (5.99)

5. Other Pre Specified Outcome: Total Activity Time (TAT)
Description: TAT is a measure of the total time that the Veteran will be participating in mini-game challenges during the 60 minute intervention session.
Time Frame: (Intervention) 2 times per week for 8 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
Minutes
  1st 5 interventions | 27.13 (2.58)
  2nd 5 interventions | 32.85 (1.9)
  3rd 5 interventions | 30.5 (2.82)

6. Other Pre Specified Outcome: Time in Therapeutic Heart Rate Range (TTR)
Description: TTR is the amount of time the Veteran spends within a target heart range of moderate to vigorous exercise prescribed as greater than 40% heart rate reserve.
Time Frame: (Intervention) 2 times per week for 8 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Xbox One Kinect Gaming
Number analyzed (Participants) | 1
Minutes
  1st 5 interventions | 48.87 (7.68)
  2nd 5 interventions | 51.20 (3.67)
  3rd 5 interventions | 38.33 (9.78)

ADVERSE EVENTS:
Time Frame: Weeks 13-21
Description: Adverse events were specifically monitored during the intervention phase (weeks 13-21). Safety was a prioritized consideration during this phase as it related to the safety and feasibility of the specific intervention. During baseline and retention phases, the participant underwent repeated assessment though was primarily under free living conditions, with no active intervention, and required minimal monitoring.
Arm/Group | Xbox One Kinect Gaming
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Small number of subjects; Potentially variable cardiovascular data due to participant lifestyle

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes